CLINICAL TRIAL: NCT05835661
Title: Nasopharyngeal Airway in Obese Patients Undergoing Painless Gastroenteroscopy Compared With Transnasopharyngeal Airway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YXLL-KY-2023(001)
Record Dates: First submitted 2023-03-28; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Complication; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — According to the preliminary results, the rate of pharyngeal pain was 20% in the transoral group and 60% in the nasal group.Bilateral test α=0.05, power=0.80, considering the 20% shedding rate, the sample size was calculated by PASS software. According to the postoperative pharyngeal pain rate, the required sample size of each group was 29, and the total sample size was 58.According to the minimum oxygen saturation in the two groups, the required sample size for each group was 123, and the total sample size was 246 cases.Since both of the two research indicators are major research indicators, it is recommended to select a larger sample size of 246 cases, which can meet the research requirements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation on the application of nasopharyngeal airway: Patients eligible for inclusion were selected, and after fully explaining the advantages and disadvantages of the two ways of nasopharyngeal airway, the patients were allowed to choose to be enrolled by themselves, and then subsequent observation was started

SUMMARY:
Painless endoscopy is a popular endoscopic diagnosis and treatment method at present, and propofol combined with fentanyl general intravenous anesthesia has been widely used in painless endoscopic diagnosis and treatment.However, the combined application of the two has an obvious respiratory center inhibition effect, leading to the decrease of blood oxygen saturation in patients, especially obese patients, more prone to blood oxygen plunge, even threatening life.Due to the potential risk of upper airway obstruction in some obese patients, intraoperative hypoventilation may occur during painless colonoscopy due to the influence of sedative and analgesic drugs, thus causing hypoxia in patients. In addition, the anatomical and pathological changes of obese patients themselves make hypoxia tolerance poor and airway establishment difficult, which may endanger the safety of patients.Currently, supracloglottic ventilation devices that have little impact on patients and are easy to accept are often used clinically to complete short daytime operations. The most common is the application of oropharyngeal ventilation to solve upper airway obstruction , however, oropharyngeal ventilation is inconvenient to use in gastroenteroscopy and treatment, while nasopharyngeal ventilation is suitable. However, based on the experience of observers,Although the nasopharyngeal airway can play a good role in the unobtrusived airway, the incidence of nasopharyngeal hemorrhage is high, and the comfort of patients is poor. Therefore, the researchers considered to directly insert the nasopharyngeal airway into the pharyngeal cavity next to the oral pad through the mouth, so as to achieve the effect of unobtrusived airway and increase the local oxygen concentration, and the idea of this experiment came from this.

DETAILED DESCRIPTION:
The purpose of this trial is to reduce complications, ensure safety during gastroenteroscopy and improve postoperative satisfaction of patients.According to the preliminary experimental results, the nasopharyngeal airway inserted by the oral pad is more convenient than the traditional operation, and the incidence of postoperative bleeding and pharyngeal pain is lower.The pros and cons of these two methods will be fully informed when the informed consent is signed with the patients at the early stage of the trial, so that the patients can voluntarily choose the implantation method.

ELIGIBILITY:
Inclusion Criteria ASA1-2; BMI≥28; Age 18-65years old

Exclusion Criteria

Pregnancy； History of allergies to propofol； history of alcohol abuse; psychiatric or neurological disorders; speech and communication disorders; auditory or visual impairments that may affect quality assessment of recovery; prior memory or cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patients are more prone to sudden drop of blood oxygen, even threatening life .Due to the potential risk of upper airway obstruction in some obese patients, intraoperative hypoventilation may occur during painless colonoscopy due to the influence of sedative and analgesic drugs, thus causing hypoxia in patients. In addition, the anatomical and pathological changes of obese patients themselves make hypoxia tolerance poor and airway establishment difficult, which may endanger the safety of patients.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Operating duration | Intraoperative (From the insertion of nasopharyngeal airway to the adjustment of position under gastroscopy)
  The period of time from the beginning of insertion of the nasopharyngeal airway until it is adjusted into place
The incidence of nasopharyngeal hemorrhage and postoperative pharyngeal pain | The whole experiment process was completed from the beginning of anesthesia induction to Forty eight hours after surgery
  The satisfaction survey was carried out in the resuscitation room after the recovery of the patients, and the adverse reactions such as bleeding and sore throat were asked

SECONDARY OUTCOMES:
The lowest drop in SPO2 during anesthesia | Intraoperative (From the beginning to the end of anesthesia)
  The lowest value of SPO2 drop during the whole operation
Postoperative satisfaction of patients | The whole experiment process was completed from the beginning of anesthesia induction to Forty eight hours after surgery
  The Minnesota satisfaction score was used for patient satisfaction. The short scale included three subscales of intrinsic satisfaction, extrinsic satisfaction and general satisfaction. The main items included: the 5-point scale was used, where 1= very dissatisfied with this aspect of my job, 2= dissatisfied with this aspect of my job;3= Not sure whether I am satisfied or dissatisfied with this aspect of my job;4= satisfied with this aspect of my job;5= Very satisfied with this aspect of my job.

CONTACTS AND LOCATIONS:
Overall Officials: ChuanYu Sun, master, Principal Investigator — Department director
Locations (1):
- YOU Qi, Jinan, China

IPD SHARING:
Plan to Share IPD: No